CLINICAL TRIAL: NCT05153018
Title: Population Immunity AgaiNst mosquitO-borne Diseases in Vanuatu
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Ministry of Health of Vanuatu (Unknown); Vanuatu National Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-100
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Arbovirus Disease; Zika; Dengue; Ross River; Chikungunya; COVID-19
Keywords: Serology; Epidemiology; Vanuatu
MeSH Terms: conditions — Zika Virus Infection; Dengue; Ross River Virus Infection; Chikungunya Fever; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A representative random sample of the population (Other): 1,200 non-febrile individuals aged older than 6 years old
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — a 4-mL blood sample collected in a dry tube

SUMMARY:
The Pacific region is facing several emerging and neglected diseases notably mosquito-borne diseases as malaria or arboviroses among which dengue, Ross River, chikungunya and Zika. These diseases are an important cause of illness and death in the Pacific and the occurrence of arboviruses has increased in the recent years. In humans, these mosquito-borne diseases often have very similar clinical presentations (an acute febrile syndrome often self-limiting). However, these infections can progress to severe and fatal prognosis.

Numerous arboviroses outbreaks and in particular dengue outbreaks have affected Vanuatu for decades. Except for DENV and Zika for which epidemiological and virological data are available for Vanuatu, the knowledge on chikungunya and Ross River circulation is very limited and needs to be defined as both viruses have intensively circulated in the region in the past. Knowledge of the level of immune protection of the population for these mosquito-borne diseases is incomplete. For this purpose, seroprevalence studies that intend to retrospectively look for antibodies (IgG) as an evidence of previous infections by a specific pathogen would be highly informative. Knowing the serological profile of the Vanuatu population for dengue and other arboviruses as Ross River, chikungunya and Zika that could have affected the country in the past would be useful in defining the population likely to be infected by future epidemics.

COVID-19 pandemic caused by SARS-CoV-2 as caused over 520 million cases since December 2019. Vanuatu has been relatively spared from the pandemic due to the establishment of a sanitary sas involving strict border control. On 04 March 2022, an active COVID-19 case was confirmed at Vila Central Hospital who had no travel history, indicating transmission at community level. Overall, a total of 8487 confirmed cases have been reported since the beginning of 2022.

Local vaccination campaign was initiated in July 2021. A seroprevalence study documenting population immunity to COVID-19 will inform of the breadth of COVID-19 epidemic in Vanuatu, contributing to the evaluation of undetected infections rate. This identification of vulnerable populations will inform local public Health strategies, including targeted vaccination campaigns.

DETAILED DESCRIPTION:
The PIANO project is a non-comparative observational prospective cross-sectional descriptive survey on a representative random sample of the population.

The study will be conducted on a 4-mL blood sample collected in a dry tube from 1,200 non-febrile individuals aged older than 6 years old.

The main objective of the current project is to determine the seroprevalence of dengue, Zika, chikungunya, Ross River and COVID-19 in Vanuatu.

ELIGIBILITY:
Inclusion Criteria:

* Individuals informed of the research and having given their written consent to participate in the study
* Individuals aged 6 years old or more
* Individuals living in Vanuatu for more than 6 months
* Individuals informed of the research, its objectives and procedure

Exclusion Criteria:

* Tourists and people present in Vanuatu for less than 6 months
* Persons intellectually disabled or under guardianship
* Persons suffering from a febrile syndrome
* Missing information related to age or hometown
* Children weighting less than 18 kg

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1122 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Determination of the seroprevalence of dengue, Zika, chikungunya, Ross River and Covid-19 in Vanuatu. | 1 year
  Exploration of vector-borne diseases seroprevalence in the main Provinces usually involved in outbreaks, the study will be implemented in the main cities of Efate, Santo, Tanna and Malekula Islands namely Port Vila, Luganville, Isangel and Lakatoro along with rural parts connected to the main city by main roads.

CONTACTS AND LOCATIONS:
Overall Officials: Myrielle Dupont-Rouzeyrol, PhD, Study Director — Institut Pasteur de Nouvelle-Calédonie
Locations (4):
- Vanuatu (4):
  - Blood centers, hospitals, health facilities, Luganville
  - Schools, Luganville
  - Blood centers, hospitals, health facilities, Port Vila
  - Schools, Port Vila